CLINICAL TRIAL: NCT01032603
Title: A Randomized Trial of Bilateral Lateral Rectus Recession Versus Unilateral Lateral Rectus Recession With Medial Rectus Resection for Intermittent Exotropia
Brief Title: Bilateral Lateral Rectus Recession Versus Unilateral Recess-Resect for Intermittent Exotropia
Acronym: IXT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Pediatric Eye Disease Investigator Group (Network); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEI-145; 2U10EY011751 (NIH)
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Exotropia
Keywords: IXT; Exotropia; Strabismus; Intermittent exotropia
MeSH Terms: conditions — Exotropia; Strabismus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bilateral lateral rectus recession (Active Comparator): Bilateral lateral rectus recession surgery
  Interventions: Procedure: Bilateral lateral rectus recession (BLRc)
- Unilateral lateral rectus recession (Active Comparator): Unilateral lateral rectus recession w/ medial rectus resection surgery
  Interventions: Procedure: Unilateral lateral rectus recession with medial rectus resection (R&R)

INTERVENTIONS:
Procedure: Bilateral lateral rectus recession (BLRc) — Bilateral lateral rectus recession surgery
  Other Names: BLR; BLRc
  Arms: Bilateral lateral rectus recession
Procedure: Unilateral lateral rectus recession with medial rectus resection (R&R) — A unilateral lateral rectus recession combined with a medial rectus resection in the same eye. Choice of eye at investigator discretion based on any interocular difference, position under anesthesia, fixation preference, or forced duction testing. Reason for choice of eye will be recorded.
  Other Names: R&R
  Arms: Unilateral lateral rectus recession

SUMMARY:
The purpose of this study is to evaluate the effectiveness of bilateral lateral rectus muscle recession versus unilateral lateral rectus recession with medial rectus resection procedures for the treatment of basic type and pseudo divergence excess type intermittent exotropia.

DETAILED DESCRIPTION:
Intermittent exotropia (IXT) is the most common form of childhood onset exotropia with an incidence of 32.1 per 100,000 in children under 19 years of age. Intermittent exotropia is characterized by an exotropia that is not constant and is mainly present when viewing at distance, but may also be present at near. Normal binocular single vision (BSV) is typically present at near when the exotropia is controlled, with evidence of normal (occasionally sub-normal) stereoacuity. Although the natural history of the condition is largely unknown, many children with IXT are treated using either surgical or non-surgical interventions. The rationale for intervention in childhood IXT is that extended periods of misalignment may lead to entrenched suppression, resulting in loss of BSV. Intervention may also aim to address the social effects caused by the appearance of misaligned eyes. Many children treated for IXT are currently treated surgically.

There is poor agreement as to which type of surgery is most effective for the correction of IXT and the debate has long been related to differentiation between IXT sub-types. Based on distance-near angle disparity, IXT sub-types are classified as: 1) basic (similar magnitude of misalignment at distance and near); 2) true divergence excess (larger at distance); 3) pseudo divergence excess (initially larger at distance, but near angle increases following occlusion or with addition of plus lenses at near); 4) convergence insufficiency (larger at near). Basic and pseudo divergence excess appear to be the most common of the sub-types, and are also the types for which there is most disagreement regarding the optimum surgical approach. The two most common procedures are bilateral lateral rectus recession (BLRrec) and unilateral lateral rectus recession combined with a medial rectus resection in the same eye (R&R). Traditionally, BLRrec has been advocated where there is a larger distance angle, and R&R where there is a similar angle at distance and near. A survey of American strabismus surgeons published in 1990 found that the majority performed BLRrec for both basic and divergence excess types. Similarly, we found by polling our investigator group that the majority still perform a BLRrec for basic type IXT. Nevertheless, controversy still exists as to which of these surgical approaches is superior. Advocates of the BLRrec procedure tend to hold that surgery should be based purely on the distance angle of deviation. Proponents of R&R surgery suggest resection of the medial rectus best addresses the exodeviation at near.

The proposed advantage of the R&R procedure is that resecting the medial rectus, with a possible longer term initial overcorrection, is necessary for a stable and superior long-term outcome. Nevertheless, those who favor the BLRrec procedure suggest that the more profound and prolonged initial overcorrection occurring with R&R is not only unnecessary, but may in fact be harmful. A persistent overcorrection may be associated with the development of diplopia, amblyopia, and loss of stereoacuity. On the other hand, critics of the BLRrec procedure suggest that long-term recurrence rates are higher. Poor motor outcomes are likely to require reoperation and therefore the long-term success rates of these surgeries have public health importance in terms of cost to society.

Evaluating initial and long-term surgical outcomes in the proposed randomized clinical trial (RCT) will answer questions regarding the failure rates of these surgeries and also provide needed data on the potential harm of each procedure.

Only one prospective randomized clinical trial addresses success rates of BLRrec versus R&R for IXT. After between 12-15 months of follow up, 82% of 17 patients undergoing an R&R had a satisfactory outcome compared to 52% of 19 patients undergoing a BLRrec. Nevertheless, there are some important limitations of this previous study. The sample size was very small. The study population was a sub-group of patients with basic type IXT, excluding patients with basic IXT whose angle of deviation increased at far distance or following occlusion, thus limiting the generalizability of the results. In addition, outcomes were assessed unmasked, potentially biasing the results. One observational study of 103 patients (90% of whom had basic type IXT) found 1-year success rates of 56% for BLRrec and 60% for R&R. A retrospective study of 115 patients with basic type IXT reported success rates of 69% for BLRrec and 77% for R&R after an average of 15 months of follow up. Other studies comparing surgery types are limited not only by retrospective study design but also by inclusion of other types of exotropia, making it difficult to interpret results. In addition, many different criteria for success are used, precluding meaningful comparison of success rates between studies. This lack of evidence makes it very difficult to counsel parents of children with IXT regarding the likely success and complication rate of either procedure, limiting our ability to make informed management decisions. Establishing the respective failure rates through the proposed study will allow physicians to offer patients the type of surgery with the highest chance of long-term success, minimizing suboptimal results and repeat surgeries.

The present study is being conducted to compare the effectiveness of BLRrec with R&R for the surgical treatment of basic type and pseudo divergence excess type IXT.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to < 11 years
* Intermittent exotropia (manifest deviation) meeting all of the following:

  * Intermittent exotropia at distance OR constant exotropia at distance and either intermittent exotropia or exophoria at near
  * Largest exodeviation at either distance, near OR remote distance between 15 and 50 prism diopters (PD) (inclusive) by prism and alternate cover test (PACT)
  * Exodeviation at least 15 PD at distance and near by PACT
  * Basic type or pseudo divergence excess type
* Stereoacuity of 400 arcsec or better at near by Preschool Randot stereotest (better of 2 measures)
* Visual acuity in the worse eye at least 0.3 logMAR (20/40 on ATS HOTV or 70 letters on E-ETDRS)
* No interocular difference of visual acuity more than 0.2 logMAR (2 lines on ATS HOTV or 10 letters on E-ETDRS testing)
* Absence of high AC/A ratio (exclude > 6:1)
* No previous intraocular surgery, strabismus surgery, or botulinum toxin treatment
* Investigator planning to perform surgery for correction of IXT
* No hyperopia greater than +3.50 D spherical equivalent (SE) in either eye

Exclusion Criteria:

* Coexisting vertical deviation, oblique muscle dysfunction, dissociated vertical deviation (DVD), or A or V pattern, any of which the investigator plans to address with vertical transposition of horizontal rectus muscles, oblique surgery, or vertical rectus muscle surgery, i.e., only small vertical deviations, oblique muscle dysfunction, DVD, and A or V patterns not requiring surgery are allowed
* Limitation of ocular rotations due to restrictive or paretic strabismus
* Craniofacial malformations affecting the orbits
* Interocular visual acuity difference of more than 0.2 logMAR (2 lines on ATS HOTV for patients 3 to < 7 years old or 10 letters on E-ETDRS for patients ≥ 7 years old) and/or investigator plans to initiate amblyopia treatment at this time.
* High AC/A ratio (exclude > 6:1 by gradient method)
* Prior strabismus surgery or botulinum toxin injection
* Ocular disorders that would reduce visual acuity (except refractive error)
* Prior intraocular or refractive surgery
* Significant neurological impairment such as cerebral palsy. Patients with mild speech and/or learning disabilities are eligible.
* Investigator planning to change refractive correction at this time (if the patient is otherwise eligible, the investigator should consider prescribing refractive correction and bringing the patient back at a later time for enrollment).

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 197 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Donahue, M.D., Ph.D., Study Chair — Pediatric Ophthalmology Service, Vanderbilt Children's Hospital, Nashville, TN
Locations (1):
- Vanderbilt Children's Hospital, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the PEDIG public website after the completion of each protocol and publication of the primary manuscript.
Time Frame: Data will be made available after publication of each primary manuscript.
Access Criteria: Users accessing the data must enter an email address.

REFERENCES:
- [Background] Repka MX, Chandler DL, Holmes JM, Donahue SP, Hoover DL, Mohney BG, Phillips PH, Stout AU, Ticho BH, Wallace DK; Pediatric Eye Disease Investigator Group. The Relationship of Age and Other Baseline Factors to Outcome of Initial Surgery for Intermittent Exotropia. Am J Ophthalmol. 2020 Apr;212:153-161. doi: 10.1016/j.ajo.2019.12.008. Epub 2019 Dec 17. PMID 31862447
- [Result] Pediatric Eye Disease Investigator Group; Writing Committee; Donahue SP, Chandler DL, Holmes JM, Arthur BW, Paysse EA, Wallace DK, Petersen DB, Melia BM, Kraker RT, Miller AM. A Randomized Trial Comparing Bilateral Lateral Rectus Recession versus Unilateral Recess and Resect for Basic-Type Intermittent Exotropia. Ophthalmology. 2019 Feb;126(2):305-317. doi: 10.1016/j.ophtha.2018.08.034. Epub 2018 Sep 3. PMID 30189281
- [Result] Holmes JM, Hercinovic A, Melia BM, Leske DA, Hatt SR, Chandler DL, Dean TW, Kraker RT, Enyedi LB, Wallace DK, Donahue SP, Cotter SA; Pediatric Eye Disease Investigator Group. Improvement in health-related quality of life following strabismus surgery for children with intermittent exotropia. J AAPOS. 2021 Apr;25(2):82.e1-82.e7. doi: 10.1016/j.jaapos.2020.11.021. Epub 2021 Apr 24. PMID 33905836
- [Result] Donahue SP, Chandler DL, Wu R, Marsh JD, Law C, Areaux RG Jr, Ghasia FF, Li Z, Kraker RT, Cotter SA, Holmes JM; Pediatric Eye Disease Investigator Group. Eight-Year Outcomes of Bilateral Lateral Rectus Recessions versus Unilateral Recession-Resection in Childhood Basic-Type Intermittent Exotropia. Ophthalmology. 2024 Jan;131(1):98-106. doi: 10.1016/j.ophtha.2023.09.004. Epub 2023 Sep 9. PMID 37696452
- [Derived] Pang Y, Gnanaraj L, Gayleard J, Han G, Hatt SR. Interventions for intermittent exotropia. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD003737. doi: 10.1002/14651858.CD003737.pub4. PMID 34516656
- See also: PEDIG Public Website — https://public.jaeb.org/pedig

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Started | 101 | 96
Completed | 86 | 77
Not Completed | 15 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession | Total
Number analyzed (Participants) | 101 | 96 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 101 | 96 | 197
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.4 (2.1) | 5.9 (1.9) | 6.2 (2.0)
Age, Customized [Count of Participants; unit: Participants]
  3 to <4 years old | 14 | 15 | 29
  4 to <5 years old | 19 | 24 | 43
  5 to <6 years old | 14 | 20 | 34
  6 to <7 years old | 15 | 10 | 25
  7 to <8 years old | 15 | 11 | 26
  8 to <9 years old | 10 | 4 | 14
  9 to <10 years old | 9 | 10 | 19
  10 to <11 years old | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 58 | 122
  Male | 37 | 38 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 58 | 55 | 113
  African American | 13 | 14 | 27
  Hispanic | 19 | 25 | 44
  Other | 11 | 2 | 13
Prior Nonsurgical Treatment [Count of Participants; unit: Participants]
  No treatment | 49 | 49 | 98
  Patching alone | 36 | 29 | 65
  Overminus spectacles alone | 6 | 4 | 10
  Vision therapy alone | 2 | 3 | 5
  Combination or other | 8 | 11 | 19
Randot Preschool Stereoacuity [Count of Participants; unit: Participants] — Stereoacuity scores (seconds of arc, or arcsec) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity.
  Participants
    40 Arcsec | 15 | 16 | 31
    60 Arcsec | 22 | 20 | 42
    100 Arcsec | 28 | 31 | 59
    200 Arcsec | 12 | 13 | 25
    400 Arcsec | 24 | 16 | 40
Randot Preschool Stereoacuity (log arcsec) [Mean (Standard Deviation); unit: logarithm of seconds of arc (log arcsec)] — Stereoacuity scores (seconds of arc) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity.
  A logarithm base 10 transformation was used to convert stereoacuity scores to the log scale to calculate descriptive statistics (reported as seconds of arc, or arcsec).
  logarithm of seconds of arc (log arcsec) | 2.1 (0.4) | 2.0 (0.3) | 2.1 (0.3)
Randot Preschool Stereoacuity (log arcsec) [Mean (Full Range); unit: logarithm of seconds of arc (log arcsec)] — Stereoacuity scores (seconds of arc) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity.
  A logarithm base 10 transformation was used to convert stereoacuity scores to the log scale to calculate descriptive statistics (reported as seconds of arc, or arcsec).
  logarithm of seconds of arc (log arcsec) | 2.1 [1.6 to 2.6] | 2.0 [1.6 to 2.6] | 2.1 [1.6 to 2.6]
Distance Randot Stereoacuity [Count of Participants; unit: Participants] — Stereoacuity scores (seconds of arc) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity.
  Participants
    60 Arcsec | 27 | 25 | 52
    100 Arcsec | 14 | 19 | 33
    200 Arcsec | 18 | 16 | 34
    400 Arcsec | 20 | 13 | 33
    Nil | 20 | 20 | 40
    Missing | 2 | 3 | 5
Distance Randot Stereoacuity (log arcsec) [Mean (Standard Deviation); unit: log arcsec] — Stereoacuity scores (seconds of arc) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity.
  A logarithm base 10 transformation was used to convert stereoacuity scores to the log scale to calculate descriptive statistics (reported as seconds of arc, or arcsec).
  log arcsec | 2.3 (0.4) | 2.3 (0.4) | 2.3 (0.4)
Distance Randot Stereoacuity (log arcsec) [Mean (Full Range); unit: log arcsec] — Stereoacuity scores (seconds of arc) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity.
  A logarithm base 10 transformation was used to convert stereoacuity scores to the log scale to calculate descriptive statistics (reported as seconds of arc, or arcsec).
  log arcsec | 2.3 [1.8 to 2.9] | 2.3 [1.8 to 2.9] | 2.3 [1.8 to 2.9]
Baseline Exotropia Magnitude by PACT at Distance [Mean (Standard Deviation); unit: Prism Diopter] — The prism and alternate cover test (PACT) is used to measure the angle of strabismus, or deviation, in prism diopters. This is measured separately at distance and at near. Smaller numbers are better because they indicate a smaller angle of deviation.
  Prism Diopter | 26 (6) | 26 (6) | 26 (6)
Baseline Exotropia Magnitude by PACT at Near [Mean (Standard Deviation); unit: Prism Diopter] — The prism and alternate cover test (PACT) is used to measure the angle of strabismus, or deviation, in prism diopters. This is measured separately at distance and at near. Smaller numbers are better because they indicate a smaller angle of deviation.
  Prism Diopter | 25 (8) | 24 (8) | 24 (8)
Baseline Exotropia Control at Distance [Mean (Standard Deviation); unit: scores on a scale] — Exotropia control was measured in points ranging from 0 to 5, with each point corresponding to the following:
  0: No exotropia unless dissociated, recovers <1 secs (phoria)
  1. No exotropia unless dissociated, recovers 1-5 secs
  2. No exotropia unless dissociated, recovers >5 secs
  3. Exotropia <50% of 30-second observation
  4. Exotropia >50% of 30-second observation
  5. Constant exotropia
  Lower scores indicate better control.
  scores on a scale | 3.4 (1.4) | 3.4 (1.2) | 3.4 (1.3)
Baseline Exotropia Control at Near [Mean (Standard Deviation); unit: scores on a scale] — Exotropia control was measured in points ranging from 0 to 5, with each point corresponding to the following:
  0: No exotropia unless dissociated, recovers <1 secs (phoria)
  1. No exotropia unless dissociated, recovers 1-5 secs
  2. No exotropia unless dissociated, recovers >5 secs
  3. Exotropia <50% of 30-second observation
  4. Exotropia >50% of 30-second observation
  5. Constant exotropia
  Lower scores indicate better control.
  scores on a scale | 1.9 (1.2) | 1.7 (1.3) | 1.8 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Suboptimal Surgical Outcome as Assessed by Motor Alignment and Stereoacuity at Near by 3 Years
Description: A participant's intermittent exotropia (IXT) was considered to be a suboptimal surgical outcome if at any visit occurring 6 months or later, ANY of the following criteria are present by masked examiner testing:
  1. Exotropia at distance OR near at any time during the exam (i.e., can be constant or intermittent; determined by a cover/uncover test) with a magnitude of ≥10Δ by SPCT, confirmed by a retest
  2. Constant esotropia at distance OR near (determined by at least 3 cover/uncover tests-one must be before any dissociation) with a magnitude of ≥6Δ by SPCT, confirmed by a retest
  3. Decrease in Randot Preschool near stereoacuity ≥2 octaves (≥0.6 log arcsec) from enrollment, or to nil, confirmed by a retest Participants who underwent reoperation (or treatment with botulinum toxin) without first meeting any of the above suboptimal surgical outcome criteria were also counted as suboptimal surgical outcomes in the primary analysis.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 101 | 96
Participants | 43 | 33
Statistical Analysis 1: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; Test type: Superiority; p = 0.24, Z test; Difference in percentage of participants = 9, 95% CI 2-sided [-6 to 23] — Proportion of participants meeting criteria was obtained by Kaplan-Meier method. BLR group=46%, RR group=37%. Probability was compared b/w groups using Z test. A group difference and 95% CI were calculated. Positive differences favor the RR group

2. Secondary Outcome: Patients With Exotropia by 3 Years
Description: Exotropia ≥10Δ by simultaneous prism and cover test (SPCT) at distance or near, confirmed by a retest, by 3 years. Criteria was met before any reoperation, and regardless of whether suboptimal surgical outcome was met by another criteria.
Time Frame: Enrollment to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 101 | 96
Participants | 31 | 22
Statistical Analysis 1: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; Test type: Superiority; p = 0.25, Z test; Difference in percentage of participants = 8, 95% CI 2-sided [-6 to 21] — Proportion of participants meeting criteria was obtained by Kaplan-Meier method. BLR group=34%, RR group=26%. Probability was compared b/w groups using Z test. A group difference and 95% CI were calculated. Positive differences favor the RR group

3. Secondary Outcome: Patients With Constant Esotropia by 3 Years
Description: Constant esotropia ≥6Δ by simultaneous prism and cover test (SPCT) at distance or near, confirmed by a retest, by 3 years. Criteria was met before any reoperation, and regardless of whether suboptimal surgical outcome was met by another criteria.
Time Frame: Enrollment to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 101 | 96
Participants | 3 | 9
Statistical Analysis 1: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; Test type: Superiority; p = 0.06, Z test; Difference in percentage of participants = -7, 95% CI 2-sided [-14 to 0.23] — Proportion of participants meeting criteria was obtained by Kaplan-Meier method. BLR group=3%, RR group=10%. Probability was compared b/w groups using Z test. A group difference and 95% CI were calculated. Positive differences favor the RR group

4. Secondary Outcome: Number of Participants With Stereo Loss by 3 Years
Description: Decrease in Preschool Randot near stereoacuity ≥2 octaves (≥0.6 log arcsec) from enrollment, or to nil, confirmed by a retest, by 3 years. Criteria was met before any reoperation, and regardless of whether suboptimal surgical outcome was met by another criteria.
Time Frame: Enrollment to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 101 | 96
Participants | 13 | 9
Statistical Analysis 1: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; Test type: Superiority; p = 0.36, Z test; Difference in percentage of participants = 4, 95% CI 2-sided [-5 to 14] — Proportion of participants meeting criteria by 3 yrs was obtained by KM method. BLR group=14%, RR group=10%. Probability was compared b/w groups using Z test. A group difference and 95% CI were calculated. Positive differences favor the RR group

5. Secondary Outcome: Number of Participants With Exotropia Control at Distance at 3 Years
Description: Exotropia control at distance was assessed in all patients who completed the 3-year visit. Numeric values for exotropia control were assigned so that the following seven categories were created:
  Not applicable (no exodeviation) (0) No exotropia unless dissociated, recovers <1 secs (phoria)
  1. No exotropia unless dissociated, recovers 1-5 secs
  2. No exotropia unless dissociated, recovers >5 secs
  3. Exotropia <50% of 30-second observation
  4. Exotropia >50% of 30-second observation
  5. Constant exotropia
Time Frame: 3 years after enrollment
Population: Includes only patients who completed the 3-year visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
Participants
  Not applicable (no exodeviation) | 19 | 25
  (0) No exotropia unless dissociated, recovers <1 s | 25 | 22
  (1) No exotropia unless dissociated, recovers 1-5 | 14 | 11
  (2) No exotropia unless dissociated, recovers >5 s | 12 | 6
  (3) Exotropia <50% of 30-second observation | 5 | 4
  (4) Exotropia >50% of 30-second observation | 6 | 4
  (5) Constant exotropia | 5 | 5

6. Secondary Outcome: Mean Distance Control at 3 Years
Description: Mean exotropia control at distance was assessed in all patients who completed the 3-year visit. All 3-year visit data will be analyzed regardless of what treatment(s) a patient has received and regardless of whether the patient has undergone reoperation. Control at distance was analyzed as a continuous variable and compared between treatment groups using analysis of covariance (ANOVA) models that adjust for the corresponding baseline value (e.g. ANCOVA model of 3-year distance control will adjust for baseline distance control).
  Numeric values for exotropia control were assigned so that the following categories were created:
  Not applicable (no exodeviation) 0: No exotropia unless dissociated, recovers <1 secs (phoria)
  1. No exotropia unless dissociated, recovers 1-5 secs
  2. No exotropia unless dissociated, recovers >5 secs
  3. Exotropia <50% of 30-second observation
  4. Exotropia >50% of 30-second observation
  5. Constant exotropia
  Lower scores indicate better control.
Time Frame: 3 years after enrollment
Population: Range of the mean was 0 to 5 for both the BLR group and for the RR group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
score on a scale | 1.2 (1.6) | 1.0 (1.6)
Statistical Analysis 1: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; 3-year control outcomes were analyzed as continuous variables and compared between treatment groups using analysis of covariance (ANOVA) models that adjust for the corresponding baseline value (e.g. ANCOVA model of 3-year distance control will adjust for baseline distance control); Test type: Superiority; p = 0.44, ANOVA

7. Secondary Outcome: Change in Distance Exotropia Control at 3 Years
Description: Change is defined as the baseline value minus the 3-year value, therefore positive change = improvement.
  Numeric values for exotropia control were assigned so that the following categories were created:
  Not applicable (no exodeviation) 0: No exotropia unless dissociated, recovers <1 secs (phoria)
  1. No exotropia unless dissociated, recovers 1-5 secs
  2. No exotropia unless dissociated, recovers >5 secs
  3. Exotropia <50% of 30-second observation
  4. Exotropia >50% of 30-second observation
  5. Constant exotropia
  Lower scores indicate better control.
Time Frame: Enrollment to 3 years
Population: Range of the mean was -3 to 5 for the BLR group and -2 to 5 for the RR group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
score on a scale | 2.3 (1.7) | 2.5 (1.7)

8. Secondary Outcome: Number of Participants With Exotropia Control at Near at 3 Years
Description: Exotropia control at near was assessed in all patients who completed the 3-year visit.
  Numeric values for exotropia control were assigned so that the following categories were created:
  Not applicable (no exodeviation) 0: No exotropia unless dissociated, recovers <1 secs (phoria)
  1. No exotropia unless dissociated, recovers 1-5 secs
  2. No exotropia unless dissociated, recovers >5 secs
  3. Exotropia <50% of 30-second observation
  4. Exotropia >50% of 30-second observation
  5. Constant exotropia
  Lower scores indicate better control.
Time Frame: 3 years after enrollment
Population: Includes only patients who completed the 3-year visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
Participants
  Not applicable (no exodeviation) | 20 | 21
  (0) No exotropia unless dissociated, recovers <1 s | 36 | 32
  (1) No exotropia unless dissociated, recovers 1-5 | 16 | 13
  (2) No exotropia unless dissociated, recovers >5 s | 6 | 4
  (3) Exotropia <50% of 30-second observation | 1 | 4
  (4) Exotropia >50% of 30-second observation | 6 | 3
  (5) Constant exotropia | 1 | 0

9. Secondary Outcome: Mean Near Control at 3 Years
Description: Mean exotropia control at near was assessed in all patients who completed the 3-year visit. All 3-year visit data will be analyzed regardless of what treatment(s) a patient has received and regardless of whether the patient has undergone reoperation. Control at near was analyzed as a continuous variable and compared between treatment groups using analysis of covariance (ANOVA) models that adjust for the corresponding baseline value (e.g. ANCOVA model of 3-year near control will adjust for baseline near control).
  Numeric values for exotropia control were assigned so that the following categories were created:
  Not applicable (no exodeviation) 0: No exotropia unless dissociated, recovers <1 secs (phoria)
  1. No exotropia unless dissociated, recovers 1-5 secs
  2. No exotropia unless dissociated, recovers >5 secs
  3. Exotropia <50% of 30-second observation
  4. Exotropia >50% of 30-second observation
  5. Constant exotropia
  Lower scores indicate better control.
Time Frame: 3 years after enrollment
Population: Range of the mean was 0 to 5 for the BLR group and 0 to 4 for the RR group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
score on a scale | 0.7 (1.2) | 0.6 (1.1)
Statistical Analysis 1: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; 3-year control outcomes were analyzed as continuous variables and compared between treatment groups using analysis of covariance (ANOVA) models that adjust for the corresponding baseline value (e.g. ANCOVA model of 3-year near control will adjust for baseline near control); Test type: Superiority; p = 0.64, ANOVA

10. Secondary Outcome: Change in Near Exotropia Control at 3 Years
Description: as for outcome 7
Time Frame: Enrollment to 3 Years
Population: Range of the mean was -3 to 4 for both the BLR and RR groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
score on a scale | 1.3 (1.6) | 1.1 (1.6)

11. Secondary Outcome: Number of Participants With Distance PACT at 3 Years
Description: The prism and alternate cover test (PACT) is used to measure the angle of strabismus, or deviation, in prism diopters. This is measured separately at distance and at near. Smaller numbers are better because they indicate a smaller angle of deviation. PACT was assessed in all patients who completed the 3-year visit.
  ∆ = prism diopters; eso = esodeviation; exo = exodeviation
Time Frame: 3 years after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
Participants
  No Deviation | 10 | 21
  1-9∆ Exo | 23 | 17
  10-14∆ Exo | 15 | 12
  15-18∆ Exo | 10 | 7
  20-25∆ Exo | 16 | 12
  30-35∆ Exo | 3 | 2
  40-45∆ Exo | 0 | 0
  10-14∆ Eso | 2 | 0
  1-9∆ Eso | 7 | 6

12. Secondary Outcome: Mean Distance PACT at 3 Years
Description: The prism and alternate cover test (PACT) is used to measure the angle of strabismus, or deviation, in prism diopters. This is measured separately at distance and at near. Smaller numbers are better because they indicate a smaller angle of deviation. Mean PACT was assessed in all patients who completed the 3-year visit. All 3-year visit data will be analyzed regardless of what treatment(s) a patient has received and regardless of whether the patient has undergone reoperation. PACT was analyzed as a continuous variable and compared between treatment groups using analysis of covariance (ANOVA) models that adjust for the corresponding baseline value (e.g. ANCOVA model of 3-year PACT at distance will adjust for baseline PACT at distance).
Time Frame: 3 years after enrollment
Population: Range of the mean was -14 to 35 for the BLR group and -6 to 30 for the RR group.
Measure: Mean (Standard Deviation); unit: prism diopters
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
prism diopters | 10 (10) | 9 (10)
Statistical Analysis 1: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; 3-year PACT outcomes were analyzed as continuous variables and compared between treatment groups using analysis of covariance (ANOVA) models that adjust for the corresponding baseline value; Test type: Superiority; p = 0.21, ANOVA

13. Secondary Outcome: Change in Distance PACT From Baseline to 3 Years
Description: The prism and alternate cover test (PACT) is used to measure the angle of strabismus, or deviation, in prism diopters. This is measured separately at distance and at near. Smaller numbers are better because they indicate a smaller angle of deviation. Change is defined as the baseline value minus the 3-year value, therefore positive change = improvement. If the 3-year PACT is an esodeviation, change in PACT from baseline is the reduction in the exodeviation plus the amount of the 3-year exodeviation.
Time Frame: Enrollment to 3 years
Population: Range of the mean was -10 to 44 for the BLR group and -5 to 36 for the RR group.
Measure: Mean (Standard Deviation); unit: prism diopters
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
prism diopters | 16 (11) | 18 (10)

14. Secondary Outcome: Number of Participants With Near PACT at 3 Years
Description: as for outcome 11
Time Frame: 3 years after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
Participants
  No Deviation | 11 | 15
  1-9∆ Exo | 21 | 24
  10-14∆ Exo | 16 | 9
  15-18∆ Exo | 11 | 5
  20-25∆ Exo | 13 | 14
  30-35∆ Exo | 3 | 3
  40-45∆ Exo | 1 | 0
  10-14∆ Eso | 1 | 0
  1-9∆ Eso | 9 | 7

15. Secondary Outcome: Mean Near PACT at 3 Years
Description: The prism and alternate cover test (PACT) is used to measure the angle of strabismus, or deviation, in prism diopters. This is measured separately at distance and at near. Smaller numbers are better because they indicate a smaller angle of deviation. Mean PACT was assessed in all patients who completed the 3-year visit. All 3-year visit data will be analyzed regardless of what treatment(s) a patient has received and regardless of whether the patient has undergone reoperation. PACT was analyzed as a continuous variable and compared between treatment groups using analysis of covariance (ANOVA) models that adjust for the corresponding baseline value (e.g. ANCOVA model of 3-year PACT at near will adjust for baseline PACT at near).
Time Frame: 3 years after enrollment
Population: Range of the mean was -14 to 40 for the BLR group and -6 to 30 for the RR group.
Measure: Mean (Standard Deviation); unit: prism diopters
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
prism diopters | 10 (11) | 9 (10)
Statistical Analysis 1: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.38, ANOVA

16. Secondary Outcome: Change in Near PACT From Baseline to 3 Years
Description: as for outcome 13
Time Frame: Enrollment to 3 years
Population: Range of the mean was -14 to 44 for the BLR group and -12 to 41 for the RR group.
Measure: Mean (Standard Deviation); unit: prism diopters
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
prism diopters | 15 (12) | 16 (12)

17. Secondary Outcome: Participants With Near Stereoacuity Measures at 3 Years
Description: Stereoacuity scores (seconds of arc) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity.
  Stereoacuity Testing: stereoacuity was assessed in current refractive correction using the following:
  Preschool Randot stereotest at near (performed at 40 cm): If stereoacuity is worse than 40 arcsec, it must be retested and the better of the 2 measurements will be used for eligibility.
  Distance Randot stereotest (performed at 3 meters)
Time Frame: 3 years after enrollment
Population: Includes only patients who completed the 3-year visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
Participants
  40 | 34 | 37
  60 | 23 | 17
  100 | 19 | 12
  200 | 3 | 4
  400 | 4 | 4
  800 | 1 | 1
  Nil | 2 | 2

18. Secondary Outcome: Mean Near Stereoacuity at 3 Years
Description: Stereoacuity scores (seconds of arc) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity.
  A logarithm base 10 transformation was used to convert stereoacuity scores to the log scale to calculate descriptive statistics (reported as seconds of arc, or arcsec).
  Stereoacuity Testing: stereoacuity was assessed in current refractive correction using the following:
  Preschool Randot stereotest at near (performed at 40 cm): If stereoacuity is worse than 40 arcsec, it must be retested and the better of the 2 measurements will be used for eligibility.
  Distance Randot stereotest (performed at 3 meters)
Time Frame: 3 years after enrollment
Population: The range of the mean was -1.6 to 3.2 for both the BLR and RR groups.
Measure: Mean (Standard Deviation); unit: logarithm of seconds of arc (log arcsec)
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
logarithm of seconds of arc (log arcsec) | 1.9 (0.3) | 1.8 (0.4)
Statistical Analysis 1: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; 3-year stereoacuity outcomes were analyzed as continuous variables and compared between treatment groups using analysis of covariance (ANOVA) models that adjust for the corresponding baseline value; Test type: Superiority; p = 0.93, ANOVA

19. Secondary Outcome: Change in Near Stereoacuity From Baseline to 3 Years
Description: Stereoacuity scores (seconds of arc) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity.
  A logarithm base 10 transformation was used to convert stereoacuity scores to the log scale to calculate descriptive statistics (reported as seconds of arc, or arcsec).
  Change is defined as the baseline value minus the 3-year value, therefore positive change = improvement.
Time Frame: Enrollment to 3 years
Population: Range of the mean was -1.3 to 1.0 for the BLR group and -1.4 to 1.0 for the RR group.
Measure: Mean (Standard Deviation); unit: logarithm of seconds of arc (log arcsec)
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
logarithm of seconds of arc (log arcsec) | 0.2 (0.4) | 0.2 (0.4)

20. Secondary Outcome: Participants Distance Stereoacuity at 3 Years
Description: as for outcome 17
Time Frame: 3 years after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
Participants
  60 | 30 | 35
  100 | 17 | 7
  200 | 20 | 14
  400 | 7 | 10
  Nil | 12 | 10
  Missing | 0 | 1

21. Secondary Outcome: Mean Distance Stereoacuity at 3 Years
Description: as for outcome 18
Time Frame: 3 years after enrollment
Population: Range of the mean was 1.8 to 2.9 for both the BLR and RR groups.
Measure: Mean (Standard Deviation); unit: logarithm of seconds of arc (log arcsec
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
logarithm of seconds of arc (log arcsec | 2.2 (0.4) | 2.2 (0.4)
Statistical Analysis 1: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p = 0.82, ANOVA

22. Secondary Outcome: Change in Distance Stereoacuity From Baseline to 3 Years
Description: as for outcome 19
Time Frame: Enrollment to 3 years
Population: Range of the mean was -0.9 to 1.1 for the BLR group and -0.8 to 1.1 for the RR group.
Measure: Mean (Standard Deviation); unit: logarithm of seconds of arc (log arcsec)
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
logarithm of seconds of arc (log arcsec) | 0.1 (0.4) | 0.1 (0.4)

23. Secondary Outcome: Health Related Quality of Life
Description: Health-related quality of life will be assessed using the Intermittent Exotropia Questionnaire (IXTQ). This questionnaire consists of 6 components:
  1. Child questionnaire - consists of 12 items which assess how the child feels about his/her eye condition.
     * One version for children aged 5 to < 8 years has a 3-level response scale
     * The version for children aged 8 years and older has a 5-level response scale
  2. Parent proxy questionnaire - consists of 12 items which assess how the parent feels the child's eye condition affects the child
  3. Parental questionnaire - consists of 17 items which assess how the child's eye condition affects the parent. Has 3 sub-scales: surgical, functional, and psycho-social.
  All scales ranged from 0 to 100; higher values indicated a better quality of life. Sub-scales were not combined, but rather were each evaluated individually on a scale of 0-100.
Time Frame: 3 years after enrollment
Population: The total number of children/patients was split between two categories: younger and older, which is why the number analyzed is different between rows. 1 patient in the BLR group and 2 patients in the RR group were missing quality of life questionnaire data. Parent information was not missing which is why the total number is equal to number analyzed
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
score on a scale
  Child 5 to 7 years old IXTQ: number analyzed (Participants) | 28 | 27
  Child 5 to 7 years old IXTQ | 91 [0 to 100] | 86 [0 to 100]
  Child 8 to 13 years old IXTQ: number analyzed (Participants) | 57 | 48
  Child 8 to 13 years old IXTQ | 82 [0 to 100] | 82 [0 to 100]
  Parent Proxy IXTQ | 86 [0 to 100] | 91 [0 to 100]
  Parent Psychosocial | 97 [0 to 100] | 100 [0 to 100]
  Parent Function | 83 [0 to 100] | 86 [0 to 100]
  Parent Surgery | 83 [0 to 100] | 92 [0 to 100]
Statistical Analysis 1: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; For the each of the two age-specific versions of the child IXTQ, the proxy questionnaire, and for each of the three parent questionnaire subscales, mean Rasch-based HRQOL scores at 3 years were compared between treatment groups using the Wilcoxon rank sum test; Test type: Superiority; p = 0.30, Wilcoxon (Mann-Whitney) — Child 5 to 7 years old
Statistical Analysis 2: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; For the each of the two age-specific versions of the child IXTQ, the proxy questionnaire, and for each of the three parent questionnaire subscales, mean Rasch-based HRQOL scores9, 10 at 3 years were compared between treatment groups using the Wilcoxon rank sum test; Test type: Superiority; p = 0.77, Wilcoxon (Mann-Whitney) — Child 8 to 13 years old
Statistical Analysis 3: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; [analysis description as in outcome 23, analysis 2]; Test type: Superiority; p = 0.51, Wilcoxon (Mann-Whitney) — Parent Proxy IXTQ
Statistical Analysis 4: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; [analysis description as in outcome 23, analysis 2]; Test type: Superiority; p = 0.42, Wilcoxon (Mann-Whitney) — Parent Psychosocial
Statistical Analysis 5: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; [analysis description as in outcome 23, analysis 2]; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney) — Parent Function
Statistical Analysis 6: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; [analysis description as in outcome 23, analysis 2]; Test type: Superiority; p = 0.64, Wilcoxon (Mann-Whitney) — Parent Surgical

24. Secondary Outcome: Cumulative Number of Patients With Reoperation by 3 Years
Description: The cumulative proportion of re-operation by 3 years was compared between treatment groups using methods similar to the primary analysis (i.e. using Kaplan-Meier method). A treatment-group difference and a corresponding 95% confidence interval were also calculated. Reasons for re-operation included:
  XT; XT and worsening stereo ; XT, worsening stereo and social concerns ; XT, diplopia, and headaches ; XT and squinting with one eye closed ; ET ; ET, worsening stereo, and diplopia; ET, worsening stereo and social concerns ; ET, worsening stereo, social concerns, and amblyopia ; Inferior oblique overaction
Time Frame: 3 years after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 101 | 96
Participants | 9 | 4
Statistical Analysis 1: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; The cumulative proportion of participants with re-operation by 3 years was obtained using the Kaplan-Meier (K-M) method. A treatment-group difference and a corresponding 95% confidence interval were calculated. Treatment-group differences were calculated as BLR minus RR; Test type: Superiority; Difference in percentage = 5, 95% CI 2-sided [-2 to 13]

25. Secondary Outcome: Number of Participants With Complete or Near-Complete Resolution at 3 Years
Description: Complete or near-complete resolution was defined as meeting all of the following at the 3 year visit: 1) exodeviation <10 Δ (tropia or phoria) by both SPCT and PACT at distance and near and ≥10 Δ reduction in PACT magnitude from the largest of the distance and near angles at enrollment, 2) esotropia <6 Δ at distance and near by SPCT, 3) no decrease in Randot Preschool stereoacuity of ≥2 octaves from the enrollment stereoacuity or to nil, 4) no reoperation or treatment with botulinum toxin, and 5) no non-surgical treatment for a recurrent or residual exodeviation.
Time Frame: 3 years after enrollment
Population: Includes only those patients that completed the 3-year visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
Participants | 26 | 35
Statistical Analysis 1: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; All treatment-group differences were calculated as the BLRc group minus the R&R group. A treatment-group difference and a corresponding 95% confidence interval were calculated; Test type: Superiority; Difference in percentage of participants = -15, 95% CI 2-sided [-30 to -.0003]

26. Secondary Outcome: Participants Suboptimal Surgical Outcome at 3 Years
Description: Suboptimal surgical outcome at the 3-year visit was defined as meeting any of the three suboptimal surgical outcome criteria at the 3-year visit (regardless of whether the criterion had been met at an earlier visit), or undergoing reoperation at any time.
  The three criteria for suboptimal surgical outcome were:
  1. Exotropia at distance OR near at any time during the exam (i.e., can be constant or intermittent; determined by a cover/uncover test) with a magnitude of ≥10Δ by SPCT, confirmed by a retest
  2. Constant esotropia at distance OR near (determined by at least 3 cover/uncover tests-one must be before any dissociation) with a magnitude of ≥6Δ by SPCT, confirmed by a retest
  3. Decrease in Randot Preschool near stereoacuity ≥2 octaves (≥0.6 log arcsec) from enrollment, or to nil, confirmed by a retest
Time Frame: 3 years after enrollment
Population: Includes only those who completed the 3 year visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
Number analyzed (Participants) | 86 | 77
Participants | 25 | 13
Statistical Analysis 1: Comparison: Bilateral Lateral Rectus Recession vs Unilateral Lateral Rectus Recession; The proportion of participants with suboptimal surgical outcome at 3 years was compared between treatment groups using Barnard's exact test, and an exact 95% CI on the treatment-group difference was calculated using Farrington-Manning scores; Test type: Superiority; Difference in percentage of participants = 12, 95% CI 2-sided [-1 to 25]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Bilateral Lateral Rectus Recession | Unilateral Lateral Rectus Recession
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/96
Other Adverse Events (participants affected / at risk) | 0/101 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT01032603/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT01032603/SAP_002.pdf
  • Informed Consent Form (2013-07-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT01032603/ICF_001.pdf